CLINICAL TRIAL: NCT05568654
Title: Reducing Antimicrobial Overuse Through Targeted Therapy for Patients With Community-Acquired Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Rothberg, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-863
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Community-Acquired Pneumonia; Antimicrobial Stewardship; Point-of-Care Testing
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: To accomplish these two aims, we will perform a, pragmatic, multicenter 2 X 2 factorial cluster randomized controlled trial with four arms:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rapid diagnostic testing (RDT) (Active Comparator): Rapid diagnostic testing: Eligible patients at hospitals randomized to this arm will undergo testing for viral pathogens (from November-April) and pneumococcal UAT and procalcitonin testing. If the patient is not being admitted to the ICU, and the patient has an admitting diagnosis of pneumonia, the form will append orders for viral testing, UAT and procalcitonin testing to providers in hospitals randomized to receive it.
  Interventions: Diagnostic Test: Rapid Diagnostic Testing
- Pharmacist-led de-escalation (Active Comparator): Pharmacist-led de-escalation: Another CDSS algorithm will identify CAP patients who meet study criteria and have negative culture results for > 48 hours and generate a list for the clinical pharmacist, who will be a member of the study team. The alerts will be audited by the pharmacist daily on weekdays at a centralized location. The pharmacist will attempt to determine whether each patient is clinically stable. The validated measures of clinical stability in patients with CAP are a) resolved vital sign abnormalities b) normal mental status c) ability to eat. If the patient appears stable, the pharmacist will communicate their recommendations for de-escalation to the clinical providers via a phone call or page.
  Interventions: Other: Pharmacist-led de-escalation
- Rapid diagnostic testing (RDT) and Pharmacist-led de-escalation (Active Comparator): Rapid diagnostic testing: Eligible patients at hospitals randomized to this arm will undergo testing for viral pathogens (from November-April) and pneumococcal UAT and procalcitonin testing. If the patient is not being admitted to the ICU, and the patient has an admitting diagnosis of pneumonia, the form will append orders for viral, UAT and procalcitonin testing to providers in hospitals randomized to receive it.
  Pharmacist-led de-escalation: Another CDSS algorithm will identify CAP patients who meet study criteria and have negative culture results for >48-hours and generate a list for the clinical pharmacist, who will be a member of the study team. The alerts will be audited by the pharmacist daily on weekdays at a centralized location. The pharmacist will attempt to determine whether each patient is clinically stable. If the patient appears stable, the pharmacist will communicate their recommendations for de-escalation to the clinical providers via a phone call or page.
  Interventions: Diagnostic Test: Rapid Diagnostic Testing; Other: Pharmacist-led de-escalation
- Usual care (no intervention) (No Intervention): Usual care

INTERVENTIONS:
Diagnostic Test: Rapid Diagnostic Testing — Eligible patients in hospitals randomized to this arm will undergo testing for viral pathogens (from November-April) and pneumococcal UAT and procalcitonin testing. A CDSS-based alert will be generated in real time. If the patient is not being admitted to the intensive care unit, the form will append orders for viral pathogen, UAT and procalcitonin testing.
  Arms: Rapid diagnostic testing (RDT); Rapid diagnostic testing (RDT) and Pharmacist-led de-escalation
Other: Pharmacist-led de-escalation — A CDSS algorithm will identify CAP patients who meet study criteria and have negative culture results for greater than 48 hours and generate a list for the antimicrobial stewardship pharmacist, who will be a member of the study team. The alerts will be audited by the pharmacist daily at a centralized location. The pharmacist will attempt to determine whether each patient is clinically stable. The validated measures of clinical stability in patients with CAP are a) resolved vital sign abnormalities (temperature, heart rate, oxygen saturation, blood pressure and respiratory rate) b) normal mental status and c) ability to eat. If the patient appears stable, the pharmacist will communicate their recommendations for de-escalation to the clinical providers via a phone call or page. The de-escalation recommendations made by the pharmacist will be based on a protocol developed by the research team.
  Arms: Pharmacist-led de-escalation; Rapid diagnostic testing (RDT) and Pharmacist-led de-escalation

SUMMARY:
The purpose of this study is to reduce the exposure of broad-spectrum antimicrobials by optimizing the rapid detection of CAP pathogens and improving rates of de-escalation following negative cultures. To accomplish this, we will perform a 3-year, pragmatic, multicenter 2 X 2 factorial cluster randomized controlled trial with four arms: a) rapid diagnostic testing b) pharmacist-led de-escalation c) rapid diagnostic testing + pharmacist-led de-escalation and d) usual care

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is a leading cause of hospitalization and inpatient antimicrobial use in the United States. However, diagnostic uncertainty at the time of initial treatment and following negative cultures is associated with prolonged exposure to broad-spectrum antimicrobials. We propose a large multicenter cluster randomized controlled trial to test two approaches to reducing the use of broad-spectrum antibiotics in adult patients with CAP a) routine use of rapid diagnostic testing at the time of admission and b) pharmacist -led de-escalation after 48 hours for clinically stable patients with negative cultures.

When a patient is admitted with a diagnosis of pneumonia, it will trigger the admission order set and if the physician is in a hospital randomized to the rapid diagnostic testing arm, a CDSS-based alert will be generated in real time, and the form will append orders for viral, UAT and procalcitonin testing. For physicians at a hospital randomized to the control condition, ordering will proceed as usual (standard-of-care). A second CDSS algorithm will identify study patients who have negative culture results (blood and/or sputum) for greater than 48 hours and generate a list for the antimicrobial stewardship pharmacist, who will be a member of the study team. The alerts will be audited by the clinical pharmacist daily on weekdays at a centralized location. In clinically stable patients from hospitals randomized to the de-escalation arm, the pharmacist will communicate their recommendations for de-escalation to the clinical providers via a phone call, Epic chat, or page. The primary outcome will be the duration of exposure to broad-spectrum antimicrobial therapy defined by the number of days of antibiotic therapy from initiation to discontinuation. Secondary outcomes will include detection of influenza/RSV, de-escalation and re-escalation to broad-spectrum antibiotics after de-escalation, total antibiotic duration, in-hospital mortality, ICU transfer after admission, healthcare-associated CDI and acute kidney injury after 48 hours.

ELIGIBILITY:
Inclusion Criteria for patient's records:

1. Men or women greater than or equal to 18 years of age
2. Admitted to a participating (i.e. enrolled and randomized) hospital
3. Admitting diagnosis of pneumonia

Exclusion Criteria:

1. Admission to intensive care unit within 24 hours of hospital admission
2. Comfort care measures only
3. Cystic fibrosis
4. Discharged from an acute care hospital in the past week
5. Patients not eligible for empiric therapy due to a known pathogen (any positive blood or respiratory cultures in the 72 hours prior to admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of days of broad-spectrum antibiotic therapy | first 21 days of admission
  duration of exposure to broad-spectrum antimicrobial therapy defined by the number of days of antibiotic therapy in the first 21 days of admission as per National Healthcare Safety Network (NHSN) guidelines

SECONDARY OUTCOMES:
viral testing ordered (yes/no) | Up to 48 hours
  Proportion of patients in whom viral testing was ordered. We will look at each virus individually as well as all viruses together (i.e. any viral testing)
detection of influenza virus (yes/no) | Up to 48 hours
  Proportion of patients who test positive for influenza
detection of RSV (yes/no) | up to 48 hours
  Proportion of patients who test positive for RSV
detection of viruses/atypical bacteria in the respiratory panel (yes/no) | up to 48 hours
  Proportion of patients who test positive for each of the viruses/atypical bacteria in the respiratory panel
treatment with anti-viral medications | up to 48 hours
  treatment with anti-viral medications (oseltamivir, zanamivir, peramivir, baloxavir, ribavirin, remdesivir, nirmatrelvir, COVID-19 medications)
treatment with antiviral medications | within 21 days
  treatment with antiviral medications (oseltamivir, zanamivir, peramivir, baloxavir, ribavirin, remdesivir, nirmatrelvir, COVID-19 medications)
S. pneumoniae urinary antigen test (UAT) performed | up to 48 hours
  Proportion of patients in whom UAT is performed
positive pneumococcal UAT | up to 48 hours
  Proportion of patients with positive pneumococcal UAT
de-escalation by 72 hours from admission (yes/no) | within 72 hours from admission.
  Proportion of patients whose broad spectrum antimicrobials (imipenem, meropenem, piperacillin-tazobactam, aztreonam, cefepime, ceftazidime, tobramycin, ceftazidime-avibactam, ceftolozane-tazobactam, meropenem-vaborbactam, imipenem-cilastatin-relebactam, cefiderocol, ceftaroline, tigecycline, eravacycline, amikacin, linezolid or vancomycin) are de-escalated
re-escalation to broad-spectrum antibiotics after de-escalation (yes/no) | by 21 days from admission
  Proportion of patients whose antibiotics were de-escalated and that were subsequently re-escalated to broad-spectrum antibiotics (imipenem, meropenem, piperacillin-tazobactam, aztreonam, cefepime, ceftazidime, tobramycin, ceftazidime-avibactam, ceftolozane-tazobactam, meropenem-vaborbactam, imipenem-cilastatin-relebactam, cefiderocol, ceftaroline, tigecycline, eravacycline, amikacin, linezolid or vancomycin).
total duration of any antibacterial antibiotic | up to 21 days
  Total duration of any antibacterial antibiotic treatment up to 21 days, including re-initiation of antibiotics
14-day mortality | up to 14 days
  proportion of patients who die by 14 days
30-day mortality | up to 30 days
  proportion of patients who die by 30 days
ICU transfer after admission (> 24 hours after admission) | up to 21 days
  proportion of patients transferred to the ICU >24 hours after admission up to 21 days
healthcare-associated C.difficile Infection (CDI) (yes/no) | after 72 hours of admission until discharge
  CDI after 72 hours of admission. Proportion of patients with CDI after 72 hours of admission (healthcare-associated CDI) until discharge
acute kidney injury after 48 hours (yes/no) after 48 hours | up to 21 days
  Proportion of patients with AKI after 48 hours of admission, up to 21 days
total inpatient cost (from hospital's cost accounting system) | from admission to discharge or 21 days, whichever comes first
  total inpatient cost (from hospital's cost accounting system) - from admission to discharge or 21 days, whichever comes first
hospital length-of-stay (days, hours) | days from the time of admission to the time of discharge
  length of stay will be calculated in days from the time of admission to the time of discharge
empyema (yes/no) | from 48 hours to 21 days
  empyema (pus in the pleural space)
30-day readmission (yes/no) | up to 30 days after discharge
  30-day hospital readmission
Infection with a resistant organism in the future (yes/no) | up to 6 months after discharge
  up to 6 months after discharge. Resistance to CAP therapy will be defined as resistance to either a respiratory quinolone or to both a beta-lactam/3rd generation cephalosporin and a macrolide. Multi-drug resistance will be defined as any CAP bacterial isolate that tests either intermediate (I) or resistant (R) to at least one agent in three or more antimicrobial classes
Procalcitonin test (PCT) performed | up to 48 hours
  Procalcitonin test (PCT) performed. Proportion of patients in whom PCT testing is performed
Procalcitonin test (PCT) values | up to 48 hours
  Procalcitonin test (PCT) values. Proportion of patients with low vs high PCT values

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rothberg, M.D., Principal Investigator — The Cleveland Clinic
Locations (12):
- United States (12):
  - Indian River Hospital, Vero Beach, Florida
  - Weston Hospital/Cleveland Clinic Florida, Weston, Florida
  - Akron General Hospital, Akron, Ohio
  - Avon Hospital, Avon, Ohio
  - Lutheran Hospital, Cleveland, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Euclid Hospital, Euclid, Ohio
  - Fairview Hospital, Fairview Park, Ohio
  - Marymount Hospital, Garfield Heights, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - Medina Hospital, Medina, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Musher DM, Thorner AR. Community-acquired pneumonia. N Engl J Med. 2014 Oct 23;371(17):1619-28. doi: 10.1056/NEJMra1312885. No abstract available. PMID 25337751
- [Background] Jain S, Self WH, Wunderink RG, Fakhran S, Balk R, Bramley AM, Reed C, Grijalva CG, Anderson EJ, Courtney DM, Chappell JD, Qi C, Hart EM, Carroll F, Trabue C, Donnelly HK, Williams DJ, Zhu Y, Arnold SR, Ampofo K, Waterer GW, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, McCullers JA, Pavia AT, Edwards KM, Finelli L; CDC EPIC Study Team. Community-Acquired Pneumonia Requiring Hospitalization among U.S. Adults. N Engl J Med. 2015 Jul 30;373(5):415-27. doi: 10.1056/NEJMoa1500245. Epub 2015 Jul 14. PMID 26172429
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Schimmel JJ, Haessler S, Imrey P, Lindenauer PK, Richter SS, Yu PC, Rothberg MB. Pneumococcal Urinary Antigen Testing in United States Hospitals: A Missed Opportunity for Antimicrobial Stewardship. Clin Infect Dis. 2020 Sep 12;71(6):1427-1434. doi: 10.1093/cid/ciz983. PMID 31587039
- [Background] Klompas M, Imrey PB, Yu PC, Rhee C, Deshpande A, Haessler S, Zilberberg MD, Rothberg MB. Respiratory viral testing and antibacterial treatment in patients hospitalized with community-acquired pneumonia. Infect Control Hosp Epidemiol. 2021 Jul;42(7):817-825. doi: 10.1017/ice.2020.1312. Epub 2020 Dec 1. PMID 33256870
- [Background] Deshpande A, Richter SS, Haessler S, Lindenauer PK, Yu PC, Zilberberg MD, Imrey PB, Higgins T, Rothberg MB. De-escalation of Empiric Antibiotics Following Negative Cultures in Hospitalized Patients With Pneumonia: Rates and Outcomes. Clin Infect Dis. 2021 Apr 26;72(8):1314-1322. doi: 10.1093/cid/ciaa212. PMID 32129438
- [Background] Madaras-Kelly K, Jones M, Remington R, Caplinger CM, Huttner B, Jones B, Samore M. Antimicrobial de-escalation of treatment for healthcare-associated pneumonia within the Veterans Healthcare Administration. J Antimicrob Chemother. 2016 Feb;71(2):539-46. doi: 10.1093/jac/dkv338. Epub 2015 Nov 3. PMID 26538501
- [Background] Higgins TL, Deshpande A, Zilberberg MD, Lindenauer PK, Imrey PB, Yu PC, Haessler SD, Richter SS, Rothberg MB. Assessment of the Accuracy of Using ICD-9 Diagnosis Codes to Identify Pneumonia Etiology in Patients Hospitalized With Pneumonia. JAMA Netw Open. 2020 Jul 1;3(7):e207750. doi: 10.1001/jamanetworkopen.2020.7750. PMID 32697323
- [Background] Haessler S, Lindenauer PK, Zilberberg MD, Imrey PB, Yu PC, Higgins T, Deshpande A, Rothberg MB. Blood Cultures Versus Respiratory Cultures: 2 Different Views of Pneumonia. Clin Infect Dis. 2020 Oct 23;71(7):1604-1612. doi: 10.1093/cid/ciz1049. PMID 31665249
- [Background] Belforti RK, Lagu T, Haessler S, Lindenauer PK, Pekow PS, Priya A, Zilberberg MD, Skiest D, Higgins TL, Stefan MS, Rothberg MB. Association Between Initial Route of Fluoroquinolone Administration and Outcomes in Patients Hospitalized for Community-acquired Pneumonia. Clin Infect Dis. 2016 Jul 1;63(1):1-9. doi: 10.1093/cid/ciw209. Epub 2016 Apr 5. PMID 27048748
- [Background] Allgaier J, Lagu T, Haessler S, Imrey PB, Deshpande A, Guo N, Rothberg MB. Risk Factors, Management, and Outcomes of Legionella Pneumonia in a Large, Nationally Representative Sample. Chest. 2021 May;159(5):1782-1792. doi: 10.1016/j.chest.2020.12.013. Epub 2020 Dec 19. PMID 33352192
- [Derived] Deshpande A, Walker R, Schulte R, Pallotta AM, Tereshchenko LG, Hu B, Kadri SS, Klompas M, Rothberg MB. Reducing antimicrobial overuse through targeted therapy for patients with community-acquired pneumonia: a study protocol for a cluster-randomized factorial controlled trial (CARE-CAP). Trials. 2023 Sep 16;24(1):595. doi: 10.1186/s13063-023-07615-3. PMID 37716990